CLINICAL TRIAL: NCT03564808
Title: Long Term Effects on Skin Hyper Pigmentation With and Without Mesenchymal Stem Cell Enriched Adipose Tissue Grafting for "Contour Deformities With Pigmentary Changes on Face"
Acronym: MSCs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCs
Record Dates: First submitted 2018-06-02; First posted 2018-06-21 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Skin Pigmentation Over Contour Deformities of Face; Trauma, Rhomberg Disease
Keywords: Contour defects, Pigmentation, Enriched fat grafting
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Quasi experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat graft enriched with MSCs (Experimental): Adipose tisse derrived MSCs
  Interventions: Drug: MSC
- Fat graft only (Experimental): Fat graft withiut enrichment with MSCs
  Interventions: Drug: MSC

INTERVENTIONS:
Drug: MSC — Adipose tissue enriched with mesenchymal stem cells

SUMMARY:
MSCs one injected along with fat, regulate pigmentation over the contour defects of face

DETAILED DESCRIPTION:
INTRODUCTION:

Contour deformities of the face requiring soft tissue augmentation are usually associated with hyper pigmentation of overlying skin. These deformities often result from a variety of conditions like trauma, infection and certain acquired diseases1. Contour deformities of face cause both functional as well as aesthetic problems for the patient. Hyper pigmentation of overlying skin makes these deformities more pronounced and iniquitous. Conventionally, contour problems are treated by using allogenic fillers, major flap surgery and fat grafting2. Flap surgery causes donor site morbidities and does not address pigmentary changes. Allogenic fillers, on the other hand,are expensive and also do not improve hyper pigmentation of overlying skin. Lasers and de-pigmentary creams have been described for addressing pigmentary issue but no satisfactory measure is available so far. Moreover, these modalities do not treat contour deformity.

Autologous fat grafting has gained acceptance to improve skin texture and post inflammatory hyper pigmentation associated with contour deformities of face2,3. Fat, being an autologous tissue, is an ideal choice to rejuvenate hyper pigmented skin owing to its abundant availability in areas like abdomen, buttocks, thighs and arms without any significant donor site morbidity. Repeat sessions of fat injection can be done if needed. Fat grafting is not new and it may be a safe and natural method to improve skin hyper pigmentation. One major problem related to fat grafting is resorption of grafted fat at recipient site ranging from 40% to 80% 4. It requires multiple sessions of fat injection. In literature, many treatment options have been utilized to solve this issue of resorption, one of these is enrichment of fat graft with mesenchymal stem cells 5. Mesenchymal stem cells derived from fatty tissue possess potential to proliferate as well as differentiate into multiple cell lines6,7. These mesenchymal cells not only increase consistency of grafted fat but also lead to rejuvenation of the skin overlying the fat grafted area and improve pigmentary changes of this overlying skin. However, previously published data has failed to establish a clear association of mesenchymal stem cells with improvement in hyper pigmentation of skin overlying fat grafted contour deformities of face. In order to find a reliable mean to decrease hyper pigmentation of skin overlying contour deformities of face, more work is needed to be done.

In the current study we propose the novel idea of lipo-filling the contour defects of face associated with overlying skin hyper pigmentation using enriched conventional fat graft with ex-vivo expanded fat derived mesenchymal stem cells to potentiate the improvement in overlying skin hyper pigmentation and to enhance reliability of the final outcome of surgery8,9,10,11.

The rationale of the study is to compare the improvement in skin hyper pigmentation after conventional fat grafting and stem cell enriched fat grafting for contour deformities of face associated with hyper pigmentation of overlying skin. If enrichment of fat graft with fat derived mesenchymal stem cells can increase its effect on improvement in the hyper pigmentation of overlying skin, this innovative strategy can render fat transfer a reliable option for soft tissue augmentation in contour deformities of face with overlying skin hyper pigmentation2. This can definitely improve final clinical outcome by decreasing donor site morbidity.

6.4 OBJECTIVES: To compare the long term effect on skin hyper pigmentation after conventional fat grafting and adipose-tissue derived mesenchymal stem cells enriched fat grafting for the treatment of deformities of the face associated with overlying skin hyper pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* contour deformities of face with pigmentary changes.

Exclusion Criteria:

* Depigmentary creams applied.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-05-25 (Estimated); Study Completion 2019-05-25 (Estimated)

PRIMARY OUTCOMES:
Pigmentary change | 6 months
  Pigmentary change will be measured by serial photographs in same specification of light and camera make and image J software 1.4 will be used to calculate image density which give objective measure of decrease in pigmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic surgery department king Edward Medical University Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No